Information letters for The Project:

Support Groups - a model for social inclusion and reduction of bullying in school



# INVITATION FOR YOUR CHILD TO PARTICIPATE IN THE RESEARCH PROJECT

"Support Groups in Schools – A Solution-Focused Approach to Inclusion and Bullying Prevention"

# Brief about the study:

- The study aims to investigate the effectiveness of Support Groups in schools to promote inclusion and prevent exclusion or bullying among students.
- Support Groups are based on a solution-focused approach, which is a method to facilitate
  change by highlighting students' strengths and resources. The initiative is based on student
  participation and initiative, aiming to promote friendship and belonging among students in
  school.
- A targeted child, in collaboration with the teacher and school nurse, selects fellow students to participate in the Support Group, but the targeted child does not participate in the group themselves.
- The study will contribute new and valuable knowledge.

# PURPOSE OF THE PROJECT AND WHY YOUR CHILD IS BEING ASKED TO PARTICIPATE

Observation studies at the primary school level in Norwegian schools have shown that students have positive experiences participating in Support Groups. However, we lack studies that measure the effectiveness of the method. At the primary school where your child is a student, we will now investigate whether Support Groups are an effective measure to increase inclusion and help students who experience exclusion or bullying. Your child has discussed with the school nurse or teacher that a Support Group might be a measure that can help them feel better at school. This is a request for your consent to allow your child to participate in a research project aimed at investigating whether Support Groups in schools are an effective measure.

### WHAT DOES THE PROJECT INVOLVE FOR YOUR CHILD?

By consenting to participate in the study, you agree that your child will answer a questionnaire that includes questions about bullying, quality of life, mental health, and a sense of mastery. The child will be asked to answer the questionnaire before the Support Group starts, after the Support Group has ended, and 3 and 6 months after the group has ended. The questionnaire also asks for information about gender, age, and who the child lives with.

It takes about 15 to 20 minutes to complete the questionnaire each time.

The questionnaire is completed while the child is at school, either on a computer or a tablet. The school nurse or teacher will be present during the completion and will be able to assist if anything is difficult or unclear. Parents/guardians have the opportunity to review the questionnaire.

# POTENTIAL BENEFITS AND DISADVANTAGES

An increasing number of students report experiencing exclusion and bullying at school. We lack knowledge about effective measures in schools that can prevent and stop bullying and increase safety and well-being among schoolchildren. Your child's participation will provide important information that will contribute to new knowledge in this area. This knowledge is important for individual children who experience bullying and exclusion, as well as for society as a whole. It is expected that your child will spend time completing the questionnaire.

# **VOLUNTARY PARTICIPATION AND RIGHT TO WITHDRAW YOUR CONSENT**

Participation in the project is voluntary. If you wish for your child to participate, you must sign the consent form on the last page. You can withdraw your consent for your child's participation at any time without giving a reason. There will be no negative consequences for you or your child if you choose not to participate or later decide to withdraw your child from the project. If you withdraw your consent, no further research will be conducted on the information about your child. You may also request access to the information stored about your child, and it will be provided within 30 days. You can also request that information in the project about your child be deleted, except where the material or information has been anonymized or published or has been included in completed analyses.

If you later wish to withdraw your consent for your child to participate or have questions about the project, you can contact the project leader (see contact information on the last page).

#### WHAT HAPPENS TO THE INFORMATION ABOUT YOUR CHILD?

The information registered about your child will only be used as described for the purpose of the project. Data collection will take place from autumn 2024 to spring 2025. The project will conclude in autumn 2028. After the research project is completed, the information about your child will be stored for five years for control purposes. Any extensions in usage and storage time can only occur after approval from REK and other relevant authorities. You have the right to access the information registered about your child and the right to correct any errors in the registered information. You also have the right to access the security measures in place for the processing of the information. You can complain about the processing of your information to the Data Protection Authority and the institution's Data Protection Officer.

- All information about your child will be handled without name and personal identification number or other directly identifiable information.
- Names and contact information will be replaced with a code stored on a separate research server, separate from other data.
- Only researchers at OsloMet will have access to identifiable personal information.
- All those handling information are bound by confidentiality, and the databases where the information is registered are handled with strict confidentiality.
- Publication of results is a necessary part of the research process. All publication will be done
  so that it will not be possible to identify your child in the results from the study when
  published. Individual participants will not be recognizable, but we are obliged to inform you
  that we cannot entirely rule out the possibility of recognition.

# **APPROVALS**

The Regional Committee for Medical and Health Research Ethics has conducted an ethical review and approved the project (Case Number: 717417). OsloMet is the responsible institution, and project leader Lisbeth Valla is responsible for data protection in the project.

We process the information based on the EU General Data Protection Regulation Article 6 No. 1a, Article 9 No. 2a, and your consent.

# **CONTACT INFORMATION**

If you have questions about the study or wish to learn more about or exercise your rights, contact: Project Leader: Lisbeth Valla: lisval@oslomet.no Phone: 96236870

Our Data Protection Officer at OsloMet can be reached via email: personvernombud@oslomet.no If you have questions related to Sikt's assessment of the project, you can contact via email: personverntjenester@sikt.no or by phone: 73 98 40 40.

# I CONSENT TO MY CHILD PARTICIPATING IN THE PROJECT AND THAT THE INFORMATION MY CHILD PROVIDES CAN BE USED AS DESCRIBED

| As a parent of (Full name), we consent to her/him that she/he participating in the project | |
|---|---|
| Place and date | Parent/guardian signature |
| | Parent/guardian name (printed) |
| Place and date | Parent/Guardian Signature |
| | Parent/Guardian Name (printed) |



# SUPPORT GROUPS IN SCHOOLS

This is a request asking if you would like to participate in a project about Support Groups in schools.

# WHY ARE YOU BEING ASKED TO PARTICIPATE?

You have talked with the school nurse or teacher about how a Support Group might help you feel



better at school. The goal of the Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. You get to choose which classmates will be in the Support Group to help. You will not participate in the Support Group yourself, but you will talk with the teacher or school nurse at school each week about how you are feeling.

We want to learn more about whether Support Groups help children who experience exclusion or bullying feel better at school. The information you provide is important for us to answer this question.

#### WHAT WILL HAPPEN IF YOU PARTICIPATE?

If you participate in the study, we will ask you to fill out a questionnaire. The questionnaire will be filled out several times during the school year, both before and after you have had a Support Group. The same questionnaire will be used each time. In the questionnaire, we ask you about whether you experience exclusion or bullying at school, how you are feeling, and how you enjoy school. It will take about 15-20 minutes to complete the questionnaire. The questionnaire will be filled out on a computer or tablet while you are at school. The school nurse or teacher will be present when you answer and can help you if anything seems difficult or unclear. All students at the school will fill out forms about how they enjoy school.

# WHAT WILL HAPPEN IF YOU DO NOT PARTICIPATE

Participation in the study is voluntary, and you can choose to withdraw at any time without giving a reason. There will be no negative consequences for you if you choose to participate. If you no longer wish to participate in the project, you can inform your parents or contact the teacher or school nurse at school. You can also contact us directly if you wish to withdraw or if you have other questions. Our phone number and email address are listed at the bottom of this page.

# **CONTACT PERSON**



# **SUPPORT GROUPS IN SCHOOLS**

This is a request asking if you would like to participate in a project about Support Groups in schools.

# **BACKGROUND AND PURPOSE**



You have discussed with the school nurse or teacher how a Support Group might help you feel better at school. The goal of the Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. You will have the opportunity to choose which classmates will be in the Support Group to help. You will not participate in the Support Group yourself, but you will talk with the teacher or school nurse at school every week about how you are feeling.

We want to learn more about whether Support Groups help children who experience exclusion or bullying feel better at school. The information you provide is important for us to answer this question.

# WHAT DOES THE STUDY INVOLVE?

If you choose to participate in the study, you will be asked to complete a questionnaire before starting the Support Group, right after the group ends, and 3 and 6 months after the group has ended. The same questionnaire will be completed each time. In the questionnaire, we will ask you questions about whether you experience exclusion or bullying at school, how you feel, and how you enjoy school.

It will take approximately 15-20 minutes to complete the questionnaire.

The questionnaire will be completed on a computer or tablet while you are at school. The school nurse or teacher will be present when you complete the questionnaire and can help you if something seems difficult or unclear. All students at the school will complete questionnaires about how they enjoy school.

# POSSIBLE BENEFITS AND DISADVANTAGES

If you choose to participate in the project, you will contribute to our understanding of whether Support Groups are an effective measure in schools for reducing bullying, increasing well-being, and improving health for all students. It is expected that you will spend time completing the questionnaire.



# WHAT HAPPENS TO THE INFORMATION ABOUT YOU?

The information we collect about you in the project will only be used to study whether Support Groups are an effective measure. All the information you provide will be kept secure, and only researchers at OsloMet will know what you have answered. The information you provide will be stored on a secure network. To ensure that no one can recognize you from your answers, we will replace your name and other identifying information with a code. It will not be possible to recognize you when the results of the project are presented.

# **PARTICIPATION**

Participation in the study is voluntary, and you can withdraw at any time without giving any reason. There will be no negative consequences for you if you choose not to participate. If you want to withdraw, you can inform your parents or contact your teacher or school nurse. You can also contact us directly if you wish to withdraw or have any other questions. Our contact information is provided at the bottom of this page.

# **CONTACT PERSON**



# INFORMATION THAT YOUR CHILD'S HEALTH INFORMATION WILL BE USED IN A RESEARCH PROJECT UNLESS YOU OPT OUT

The Regional Committee for Medical and Health Research Ethics (REK) has approved the research project "Support Groups in Schools – A Solution-Focused Approach to Inclusion and Bullying Prevention." REK has granted an exemption from the rule of obtaining active consent, but you have the right to decide that your child will not participate. If you do not want information about your child to be used in the project, you must actively opt out of your child's participation within 4 weeks.

# WHY WE WANT TO USE YOUR CHILD'S HEALTH INFORMATION

The purpose of the research project is to investigate the effect of Support Groups in schools among students in 5th to 7th grade. Support Groups are a measure based on student participation and initiative, using a solution-focused methodology aimed at preventing bullying and promoting friendship and belonging among students in school. The school where your child is a student has agreed to participate in the project. All students in 5th to 7th grade at the school are invited to participate in the project. Your child is not directly involved in a Support Group but is a student at a school that uses Support Groups as a measure. To ensure the study's greatest value, it is important that as many students as possible participate.

# WHAT DOES PARTICIPATION MEAN FOR YOUR CHILD?

In the project, we will collect and register information about your child. We will gather relevant information by asking your child to complete a questionnaire. The questionnaire will be completed four times during the school year. The questionnaire will include questions from the annual student survey, which in this project will be used for research. In the student survey, students will answer questions about whether they have experienced bullying, how they enjoy school, whether they look forward to going to school, and if they feel safe at school. The questionnaire is answered anonymously, and it will not be possible to recognize your child's answers in the results.

The survey will take 15-20 minutes to complete each time. It will be completed on a computer or tablet in the classroom with a teacher or school nurse present. The teacher or school nurse can help if your child finds the questions difficult to understand or answer. There is a low risk that your child will experience discomfort, burden, or harm by answering the survey.

It may be relevant to establish Support Groups for students who experience exclusion and bullying. If this becomes relevant for your child, you will be contacted by the teacher or school nurse. You will then receive a separate information letter explaining what participation entails and will be asked for written consent for your child to participate in the research project.

#### **VOLUNTARY PARTICIPATION**

If you accept that your child's health information is used as described above, you do not need to take any action.

If you do not accept that your child's health information is used as described above, you must opt out within four weeks.

You can do this by calling, sending an email or SMS, or filling out the response slip on the last page and sending it to the specified address. Please see the section on contact information.

If you do not opt out now, you can still opt out later at any time without giving any reason.

There will be no negative consequences for you or your child if you choose not to participate or later decide to withdraw. If you later decide to withdraw your participation, we will not continue to collect further information about your child.

#### WHAT HAPPENS TO YOUR CHILD'S INFORMATION?

All information registered about your child is anonymous, and it will not be possible for researchers, school staff, or in the study's published results to identify your child.

The information registered about your child will only be used as described in this letter. The project will end in 2028. The information about your child will be stored for five years after the project ends for control purposes. Any extensions in usage and storage time can only occur after approval from REK and other relevant authorities. You also have the right to access the security measures for the processing of the information.

# **CONTACT INFORMATION**

If you have any questions about the study or wish to learn more about or exercise your rights, please contact: Project Leader: Lisbeth Valla: lisval@oslomet.no Phone: 96236870

Our Data Protection Officer at OsloMet, can be reached via email: <a href="mailto:personvernombud@oslomet.no">personvernombud@oslomet.no</a>

If you have questions related to Sikt's assessment of the project, you can contact via email: personverntjenester@sikt.no or by phone: 73 98 40 40.

# I DO $\underline{\mathsf{NOT}}$ WANT MY CHILD'S INFORMATION TO BE USED IN THE RESEARCH PROJECT

| | of participation in research, please contact the project manager via ou can also fill out this response slip and submit. |
|---|---|
| Place and date | Your signature |
| Your name in canital | etters |



# INFORMATION THAT YOUR CHILD'S HEALTH INFORMATION WILL BE USED IN A RESEARCH PROJECT UNLESS YOU OPT OUT

The Regional Committee for Medical and Health Research Ethics (REK) has approved the research project "Support Groups in Schools" – REK has granted an exemption from the rule of obtaining active consent, but you have the right to decide that your child will not participate. If you do not want information about your child to be used in the project, you must actively opt out of your child's participation within 4 weeks.

#### WHY WE WANT TO USE YOUR CHILD'S HEALTH INFORMATION

The school where your child is a student has agreed to participate in a research project. Your child's school has not implemented the "Support Groups" measure but will participate as a control school in the project. The purpose of the project is to investigate whether the measure has an effect on reducing bullying and increasing well-being in school. All students in 5th to 7th grade at the school are invited to participate in the project. For the study to have the greatest possible value, it is important that as many students as possible participate.

# WHAT DOES PARTICIPATION INVOLVE FOR YOUR CHILD?

In the project, we will collect and register information about your child. We will gather relevant information by asking your child to complete a questionnaire. The questionnaire will be completed four times during the school year. The questionnaire will include questions from the annual student survey, which in this project will be used for research. In the student survey, students will answer questions about whether they have experienced bullying, how they enjoy school, whether they look forward to going to school, and if they feel safe at school. The questionnaire is answered anonymously, and it will not be possible to recognize your child's answers in the results.

The survey will take 15-20 minutes to complete each time. It will be completed on a computer or tablet in the classroom with a teacher or school nurse present. The teacher or school nurse can help if your child finds the questions difficult to understand or answer. There is a low risk that your child will experience discomfort, burden, or harm by answering the survey.

### **VOLUNTARY PARTICIPATION**

If you accept that your child's health information is used as described above, you do not need to take any action.

If you do not accept that your child's health information is used as described above, you must opt out within four weeks. You can do this by calling, sending an email or SMS, or filling out the

response slip on the last page and sending it to the specified address. Please see the section on contact information.

If you do not opt out now, you can still opt out later at any time without giving any reason. There will be no negative consequences for you or your child if you choose not to participate or later decide to withdraw. If you later decide to withdraw your participation, we will not continue to collect further information about your child.

# WHAT HAPPENS TO YOUR CHILD'S INFORMATION?

All information registered about your child is anonymous, and it will not be possible for researchers, school staff, or in the study's published results to identify your child.

The information registered about your child will only be used as described in this letter. The project will end in 2028. The information about your child will be stored for five years after the project ends for control purposes. Any extensions in usage and storage time can only occur after approval from REK and other relevant authorities. You also have the right to access the security measures for the processing of the information.

#### **CONTACT INFORMATION**

If you have any questions about the study or wish to learn more about or exercise your rights, please contact: Project Leader: Lisbeth Valla: lisval@oslomet.no Phone: 96236870

Our Data Protection Officer at OsloMet, can be reached via email: <a href="mailto:personvernombud@oslomet.no">personvernombud@oslomet.no</a>

If you have questions related to Sikt's assessment of the project, you can contact via email: personverntjenester@sikt.no or by phone: 73 98 40 40.

# I DO $\underline{\mathsf{NOT}}$ WANT MY CHILD'S INFORMATION TO BE USED IN THE RESEARCH PROJECT

| • | of participation in research, please contact the project manager via ou can also fill out this response slip and submit. |
|---|---|
| Place and date | Your signature |
| Your name in canital le | etters |



# SUPPORT GROUPS IN SCHOOLS

This is a request asking if you would like to participate in a project about Support Groups in schools.

#### **BACKGROUND AND PURPOSE**



The school where you are a student is participating in a research project about Support Groups in schools. The goal of a Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. We want to learn more about Support Groups, and the information you provide is important for us to answer this question.

# WHAT DOES THE STUDY INVOLVE?

If you choose to participate in the study, you will be asked to complete the student survey both before the school starts with the Support Group and after the project is finished. We will also ask you to complete some of the questions from the student survey at two additional time points (4 months after the project starts and 6 months after the project ends). In the questionnaire, we will ask you questions about whether you experience exclusion or bullying at school, how you are feeling, and how you enjoy school.

It will take about 15-20 minutes to complete the questionnaire each time.

The questionnaire will be completed on a computer or tablet while you are at school. The school nurse or teacher will be present when you complete the questionnaire and will be able to help you if something seems difficult or unclear. All students in 5th to 7th grade at the school will complete the same questionnaire.

### **POSSIBLE BENEFITS AND DISADVANTAGES**

If you choose to participate in the project, you will help us gain more knowledge about whether Support Groups are a useful measure in schools for reducing bullying and increasing well-being and health for all students. It is expected that you will spend time completing the questionnaire.

# WHAT HAPPENS TO THE INFORMATION ABOUT YOU?

The information we collect about you in the project will only be used to study whether Support Groups are a useful measure. All the information you provide will be kept secure. The questionnaire is answered anonymously, and it will not be possible to recognize your answers in the results.



# **PARTICIPATION**

Participation in the study is voluntary, and you can withdraw at any time without giving any reason. There will be no negative consequences for you if you choose not to participate. If you wish to withdraw, you can inform your parents or contact your teacher or school nurse. You can also contact us directly if you want to withdraw or have any other questions. Our contact information is provided at the bottom of this page.

# **CONTACT PERSON**



# QUESTION ABOUT PARTICIPATION IN A RESEARCH PROJECT

This is a request asking if you would like to participate in a research project.

# **Background and Purpose**



The school where you are a student is participating in a research project about Support Groups in schools. Your school has not yet implemented Support Groups but is a control school in the project. Many students experience exclusion or bullying, and the purpose of the research project is to gain knowledge about measures in schools that can help students feel better. We want to learn more about Support Groups, and the information you provide is important for us to answer this question.

#### WHAT DOES THE STUDY INVOLVE?

If you choose to participate in the study, you will be asked to complete the student survey at several points, both before the project starts and after it has ended. In addition, we will ask you to complete some of the questions from the student survey at two time points (4 months after the project starts and 6 months after it ends). In the questionnaire, we will ask you about whether you experience exclusion or bullying at school, how you are feeling, and how you enjoy school.

It will take about 15-20 minutes to complete the questionnaire each time. The questionnaire will be completed on a computer or tablet while you are at school. The school nurse or teacher will be present when you complete the questionnaire and can help you if something seems difficult or unclear.

All students in grades 5-7 at the school will complete the same questionnaire.

# **POSSIBLE BENEFITS AND DISADVANTAGES**

If you choose to participate in the project, you will help us gain more knowledge about whether Support Groups are a useful measure in schools for reducing bullying and increasing well-being and health for all students. It is expected that you will spend time completing the questionnaire.

#### WHAT HAPPENS TO THE INFORMATION ABOUT YOU?

The information we collect about you in the project will only be used to study whether Support Groups are a useful measure. All the information you provide will be kept secure. The questionnaire is answered anonymously, and it will not be possible to recognize your answers in the results.



# **PARTICIPATION**

Participation in the study is voluntary, and you can withdraw at any time without giving any reason. There will be no negative consequences for you if you choose not to participate. If you want to withdraw, you can inform your parents or contact your teacher or school nurse. You can also contact us directly if you want to withdraw or have any other questions. Our contact information is provided at the bottom of this page.

# **CONTACT PERSON**



# INVITATION FOR YOUR CHILD TO PARTICIPATE IN THE RESEARCH PROJECT

# "Support Groups in Schools – A Solution-Focused Approach to Inclusion and Bullying Prevention"

**Brief about the study:** The study aims to investigate the effect of Support Groups in schools to promote inclusion and prevent exclusion or bullying among students. Support Groups are based on a solution-focused approach, which is a method to facilitate change by highlighting students' strengths and resources. The initiative is based on student participation and initiative, aiming to promote friendship and belonging among students in school.

The study will contribute new and valuable knowledge.

# PURPOSE OF THE PROJECT AND WHY YOUR CHILD IS BEING ASKED TO PARTICIPATE

Observation studies at the primary school level in Norwegian schools have shown that students have positive experiences participating in Support Groups. At the primary school where your child is a student, we are now investigating whether Support Groups are an effective measure to increase inclusion and help students who experience exclusion or bullying. Your child has participated in a Support Group as a peer. Peers help other students feel better at school through activities that can promote friendship and inclusion. We want to gather more information about what it is like to be a peer. Therefore, we are asking for your consent for your child to participate in the research project.

# WHAT DOES THE PROJECT INVOLVE FOR YOUR CHILD?

By consenting to participate in the study, you agree that we can interview your child after a Support Group has been conducted. The interview will take about 1 hour, and we will ask your child about their experiences as a peer and how they contributed to helping other students feel better at school. When the conversation is over, a school nurse or teacher will be present in case your child feels the need to talk more. Parents/guardians have the opportunity to review the interview guide before the conversation takes place.

#### POSSIBLE BENEFITS AND DISADVANTAGES

An increasing number of students report experiencing exclusion and bullying in school. We lack knowledge about effective measures in schools that can prevent and stop bullying and increase safety and well-being among schoolchildren. Your child's participation will provide important information that will contribute to new knowledge in this area. This knowledge is important for individual children who experience bullying and exclusion, as well as for society as a whole. It is expected that your child will spend time participating in the interview.

# **VOLUNTARY PARTICIPATION AND THE POSSIBILITY TO WITHDRAW YOUR CONSENT**

Participation in the project is voluntary. If you want your child to participate, you sign the consent form on the last page. You can withdraw your consent for your child's participation at any time without giving a reason. There will be no negative consequences for you or your child if you choose not to participate or later decide to withdraw your child from the project. If you withdraw your consent, no further research will be conducted on the information about your child. You may also request access to the information stored about your child, and it will be provided within 30 days. You can also request that information in the project about your child be deleted, except where the material or information has been anonymized or published or has been included in completed analyses.

If you later wish to withdraw your consent for your child to participate or have questions about the project, you can contact the project leader (see contact information on the last page).

#### WHAT HAPPENS TO THE INFORMATION ABOUT YOUR CHILD?

The information registered about your child will only be used as described for the purpose of the project. Data collection will take place from autumn 2024 to spring 2025. The project will conclude in autumn 2028. After the research project is completed, the information about your child will be stored for five years for control purposes. Any extensions in usage and storage time can only occur after approval from REK and other relevant authorities. You have the right to access the information registered about your child and the right to correct any errors in the registered information. You also have the right to access the security measures in place for the processing of the information. You can complain about the processing of your information to the Data Protection Authority and the institution's Data Protection Officer.

- All information about your child will be handled without name and personal identification number or other directly identifiable information.
- Names and contact information will be replaced with a code stored on a separate research server, separate from other data.
- Only researchers at OsloMet will have access to identifiable personal information.
- All those handling information are bound by confidentiality, and the databases where the information is registered are handled with strict confidentiality.
- Publication of results is a necessary part of the research process. All publication will be done
  so that it will not be possible to identify your child in the results from the study when
  published. Individual participants will not be recognizable, but we are obliged to inform you
  that we cannot entirely rule out the possibility of recognition.

# **APPROVALS**

The Regional Committee for Medical and Health Research Ethics has conducted an ethical review and approved the project (Case Number: 717417). OsloMet is the responsible institution, and project leader Lisbeth Valla is responsible for data protection in the project. We process the information based on the EU General Data Protection Regulation Article 6 No. 1a, Article 9 No. 2a, and your consent.

# **CONTACT INFORMATION**

If you have questions about the study or wish to learn more about or exercise your rights, contact: Project Leader: Lisbeth Valla: lisval@oslomet.no Phone: 96236870

Our Data Protection Officer at OsloMet can be reached via email: personernombud@oslomet.no If you have questions related to Sikt's assessment of the project, you can contact via email: personverntjenester@sikt.no or by phone: 73 98 40 40.

# I AGREE THAT MY CHILD CAN PARTICIPATE IN THE PROJECT AND THAT THE INFORMATION MY CHILD PROVIDES CAN BE USED AS DESCRIBED

| As parents of (Full name), we consent to her/him participating in the project | |
|---|---|
| Place and date | Parent/Guardian signature |
| | Parent/Guardian name (printed) |
| Place and date | Parent/Guardian signature |
| | Parent/Guardian Name (printed) |



# SUPPORT GROUPS IN SCHOOLS

This is a request asking if you would like to participate in a project about Support Groups in schools.

#### WHY ARE YOU BEING ASKED TO PARTICIPATE?



You have participated as a peer in a Support Group at your school, and we would like to hear from you about your experience as a peer in such a group. The goal of the Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. We want to learn more about Support Groups and what it is like to be a peer. Information from you is important for us to get answers to these questions.

# WHAT WILL HAPPEN IF YOU PARTICIPATE?

If you decide to participate in the study, we would like to talk to you after your participation in a Support Group. We will ask you about your experiences and what it was like to be a peer in a Support Group. The conversation will take about one school hour, and it will be recorded to help us better remember what you tell us. Everything you say will be anonymous, and your name will not appear in anything you tell us. When the conversation is over, a school nurse or teacher at your school will be present in case you feel the need to talk more.

# WHAT WILL HAPPEN IF YOU DO NOT PARTICIPATE?

Participation in the study is voluntary, and you can decide at any time that you no longer wish to participate without giving any reason. There will be no negative consequences for you if you choose not to participate. If you no longer wish to participate in the project, you can inform your parents or contact a teacher or school nurse at the school. You can also contact us directly if you want to withdraw or have other questions. You can find our phone number and email address at the bottom of this page.

# **CONTACT PERSON**



# SUPPORT GROUPS IN SCHOOLS

This is a request asking if you would like to participate in a project about Support Groups in schools.

#### WHY ARE YOU BEING ASKED TO PARTICIPATE?



You have participated as a peer in a Support Group at your school, and we would like to hear from you about your experience as a peer in such a group. The goal of the Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. We want to learn more about Support Groups and how it feels to be a peer. Information from you is important for us to get answers to these questions.

# WHAT WILL HAPPEN IF YOU PARTICIPATE?

If you decide to participate in the study, we would like to talk to you after the Support Group has been conducted. We will ask you about your experiences and what it was like to be a peer in a Support Group. The conversation will take about one school hour, and it will be recorded to help us better remember what you tell us. Everything you say will be anonymous, and your name will not appear in anything you tell us. When the conversation is over, a school nurse or teacher at your school will be present in case you feel the need to talk more.

### WHAT WILL HAPPEN IF YOU DO NOT PARTICIPATE?

Participation in the study is voluntary, and you can decide at any time that you no longer wish to participate without giving any reason. There will be no negative consequences for you if you choose not to participate. If you no longer wish to participate in the project, you can inform your parents or contact a teacher or school nurse at the school. You can also contact us directly if you want to withdraw or have other questions. You can find our phone number and email address at the bottom of this page.

#### **CONTACT PERSON**



# SUPPORT GROUPS IN SCHOOLS

This is a request asking if you would like to participate in the research project "Support Groups in Schools."

#### **BACKGROUND AND PURPOSE**

You are a school nurse or teacher at a school participating in the research project on Support Groups in Schools. The goal of the Support Group is to help students who experience exclusion or bullying feel better at school through support and help from fellow students. The purpose of the research project is to investigate whether Support Groups are an effective measure in schools to reduce bullying and increase well-being among students. As part of the project, we also want to gather more information about the experiences of teachers or school nurses in implementing the Support Groups in schools. Your information is important for us to answer this question.

### WHAT DOES THE STUDY INVOLVE?

If you choose to participate in the study, you will be interviewed after you have conducted one or more Support Groups. We will ask you about your experiences with conducting such a group. The interview will last about 1 hour and will be recorded.

# **POSSIBLE BENEFITS AND DISADVANTAGES**

If you choose to participate in the project, you will contribute to our knowledge about the implementation of Support Groups as a measure in schools to reduce bullying and increase well-being and health for all students. It is expected that you will set aside time for the interview.

# WHAT HAPPENS TO THE INFORMATION ABOUT YOU?

The information we collect about you in the project will only be used to study whether Support Groups are a useful measure. All the information you provide will be securely stored, and only researchers at OsloMet will know what you have answered. The information from you will be stored on a secure network. To ensure that no one can recognize you from the information you provide, we will replace your name and other identifying details with a code. It will not be possible to recognize you when the results from the project are presented.

# **PARTICIPATION**

Participation in the study is voluntary, and you can withdraw at any time without giving any reason. There will be no negative consequences for you if you choose not to participate. If you wish to withdraw or have any other questions about the project, you can contact us directly. Our contact information is at the bottom of this page.



| CONTACT PERSON | |
|---|---|
| Lisbeth Valla, tel 96236870 | email, <u>lisval@oslomet.no</u> |
| . ACREE TO THE BROAFST | AND THAT THE INFORMATION I PROVIDE MAY BE USED AS |
| DESCRIBED | AND THAT THE INFORMATION I PROVIDE MAY BE USED AS |
| (Full name) we agree to particip | pata in the project |
| (ruii name) we agree to particip | iate in the project |
| Place and date | <u>signature</u> |